CLINICAL TRIAL: NCT00182897
Title: Providers and Alzheimer's Caregivers Together
Brief Title: PACT: Providers and Alzheimer's Caregivers Together
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IA0081; 5R01AG016328 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2006-11

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: caregiver; home health care; coping
MeSH Terms: conditions — Alzheimer Disease; Dementia

INTERVENTIONS:
Behavioral: Skills Building for Caregiver Health and Care-recipient

SUMMARY:
The primary goal of the study is documentation of effectiveness of a home-based intervention to reduce caregiver burden related to dementia caregiving, improve caregiver health status, and reduce caregiver and care recipient resource utilization.

DETAILED DESCRIPTION:
This study focuses on an underserved, understudied population: African American and White homebound persons with dementia and their caregivers (CGs). Severe dementia, frailty, multiple disabling co-morbid diseases, lack of transportation, inability to afford or obtain a sitter for the care recipient (CR), and lack of time in a CG's burdened daily schedule may prevent care dyads (caregivers and their family member with dementia) from receiving services in primary care settings and from participating in clinical studies. Homebound issues may be particularly important for African American CGs, yet the minority CG literature has not addressed relevant issues for homebound dyads. Nor are the chronic needs of homebound dementia care dyads adequately attended by the current home health care system, which now focuses on skilled nursing care. This study has been designed to address these research deficits. The study will examine the benefit (through improving depression, anxiety, and health perception) and the cost-effectiveness of home-based dementia caregiving interventions, with attention to both the informal care provided by the CG and the use of formal care services.

Care dyads will be randomized to either Usual Care or Enhanced Care. Both Usual Care and Enhanced Care caregivers will receive usual home health care delivered by home health nurses on the schedule determined by the patient's needs and set by the home care agency. For the Enhanced Care caregivers, to ensure protocol adherence, using the same schedule as the home health visits, trained interventionists from the research staff will deliver the intervention. The interventionists will teach dementia family caregivers to cope with difficult care recipient behaviors and challenges to caregiving and will teach caregivers how to cope with their own responses to caregiving. Following established protocols and using fifth grade level pamphlets and educational material, the interventionists will tailor the intervention sessions to meet the individual needs of each care dyad in their own home environment. Enhanced Care sessions will not exceed 60 minutes. Research specialists will perform data collection visits in the care dyads' homes at baseline, within 2 weeks of home care ending and six months.

ELIGIBILITY:
Inclusion Criteria:

Care Recipient - Inclusion Criteria (must have all)

* Documented diagnosis of dementia or Mini-Mental State Exam score <23
* Functional impairment: presence of two IADL (Instrumental Activities of Daily Living) impairment (transportation, shopping) or one Activities of Daily Living (ADL) impairment (bathing, toileting)

Caregiver - Inclusion Criteria (must have all)

* At least 21 years old
* A family member of the care recipient
* Must have a telephone
* Must plan to remain in the area for the duration of the intervention and follow-up
* Must have been a caregiver for more than 6 months
* Must provide at least 4 hours of supervision or direct assistance per day for the care recipient

Exclusion Criteria:

Care Recipient

* Any terminal illness with life expectancy of less than 6 months
* Active treatment (chemotherapy or radiation therapy) for cancer
* More than three acute medical hospitalizations in the past year (other than psychiatric or Alzheimer's Disease related admissions)
* Schizophrenia
* Dementia secondary to head trauma
* Blindness or deafness if either disability prohibits them from data collection or participation in the interventions

Caregiver

* Any terminal illness with life expectancy of less than 6 months
* Active treatment (chemotherapy or radiation therapy) for cancer
* More than three acute medical hospitalizations in the past year
* Imminent placement of care recipient into a nursing home (within 6 months)
* Involvement in another clinical trial for caregivers, including REACH
* Miscellaneous barriers such as transportation, commitment, hesitancy, etc.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2000-10; Study Completion 2005-11

PRIMARY OUTCOMES:
General well-being, measured with the revised Rand General Well-Being Scale
caregiver's level of distress with care recipient behaviors, measured with the Revised Memory and Behavior Problems Checklist at Baseline, within 2 weeks of home care ending and six months.

SECONDARY OUTCOMES:
Determine the cost-effectiveness of home-based intervention; data will be collected at Baseline, within 2 weeks of home care ending and six months.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Nichols, PhD, Principal Investigator — Program Director, Interprofessional Team Training & Development, Veterans Affairs Medical Center; Associate Professor, Preventive Medicine and Medicine, University of Tennessee Health Science Center
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

REFERENCES:
- [Background] Burns R, Nichols LO, Martindale-Adams J, Graney MJ, Lummus A. Primary care interventions for dementia caregivers: 2-year outcomes from the REACH study. Gerontologist. 2003 Aug;43(4):547-55. doi: 10.1093/geront/43.4.547. PMID 12937333
- [Background] Connell CM, Gibson GD. Racial, ethnic, and cultural differences in dementia caregiving: review and analysis. Gerontologist. 1997 Jun;37(3):355-64. doi: 10.1093/geront/37.3.355. PMID 9203759
- [Background] Haley WE, Roth DL, Coleton MI, Ford GR, West CA, Collins RP, Isobe TL. Appraisal, coping, and social support as mediators of well-being in black and white family caregivers of patients with Alzheimer's disease. J Consult Clin Psychol. 1996 Feb;64(1):121-9. doi: 10.1037//0022-006x.64.1.121. PMID 8907091
- [Background] Hall GR, Buckwalter KC, Stolley JM, Gerdner LA, Garand L, Ridgeway S, Crump S. Standardized care plan. Managing Alzheimer's patients at home. J Gerontol Nurs. 1995 Jan;21(1):37-47. doi: 10.3928/0098-9134-19950101-08. PMID 7852717